CLINICAL TRIAL: NCT06238778
Title: A Phase 2b Randomized, Double-blind Trial Comparing HDV-Insulin Lispro Versus Insulin Lispro Alone in Adults With Type 1 Diabetes Receiving Insulin Degludec
Brief Title: Phase 2b Trial Comparing HDV-Insulin Lispro to Insulin Lispro in Adults With Type 1 Diabetes Receiving Insulin Degludec
Acronym: OPTI-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diasome Pharmaceuticlas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP 01-2023-01
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus Type 1; CGM; Randomized; HDV; Lispro
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Randomized, double blind interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Enrolled subjects randomized to either the treatment arm or the control arm. The patient, the study site personnel, the CRO, and the sponsor are blinded to which group the patient is randomized to. Only the site pharmacist, and one study monitor from the CRO are unblinded. The Medical Monitor is blinded unless there is a medical reason for unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HDV Lispro (HDV-L) (Experimental): Subjects in this arm will use degludec as their daily basal insulin, and HDV-lispro as their bolus insulin
  Interventions: Drug: HDV-Lispro
- Lispro (LIS) (Active Comparator): Subjects in this arm will use degludec as their daily basal insulin and lispro as their bolus insulin
  Interventions: Drug: Lispro

INTERVENTIONS:
Drug: HDV-Lispro — HDV-L will be used as the mealtime insulin
  Other Names: HDV-L
  Arms: HDV Lispro (HDV-L)
Drug: Lispro — Lispro will be used as the mealtime insulin
  Other Names: LIS
  Arms: Lispro (LIS)

SUMMARY:
The goal of this study is to see if directing insulin to the liver will improve the low blood sugar that sometimes happens when injecting insulin in Type 1 diabetes patients. Participants will use continuous glucose monitoring to measure the sugar levels in their blood, and work with the doctor to find the best doses. One group of patients will get the liver targeting insulin, and the other group will use insulin they normally use for treating Type 1 diabetes. The participant will be part of the study for up to 32 weeks.

DETAILED DESCRIPTION:
Individuals age 18 up to 80 years with Type 1 diabetes using multiple daily injections of bolus insulin plus basal insulin will be enrolled into a double-blind randomized controlled trial to assess the efficacy, safety, and tolerability of Hepatocyte-Directed Vesicles-insulin lispro (HDV-L) versus lispro alone (LIS) used in combination with insulin degludec. The study includes (1), a screening period up to 3 weeks, (2), a Run-in Period of 2 weeks to assess eligibility and to transition to use of insulin lispro and insulin degludec and unmasked continuous glucose monitoring (CGM), )3), a 12-week dose optimization period to optimize bolus and basal insulin doses,, (4), a 13-week maintenance period, and (5), a 2 -week transition follow-up period.

The primary objective of the study is to determine if the addition of HDV to insulin lispro results in an improvement in glycemic control as defined by decreasing evidence of nocturnal hypoglycemia while maintaining or improving glycated hemoglobin (HbA1c). Other outcomes related to glycemic control will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis Type 1 diabetes with C-peptide <=0.6 ng/mL and using insulin for at least 6 months
* willing to use study provided insulin as the only bolus insulin and insulin degludec as the basal insulin
* willing to use CGM device throughout the study
* screening A1C >= 6.5% and <= 10.0% daily insulin dose <= 1.25 U/kg/day

Exclusion Criteria:

* known or specific allergy to any component of the study drug, the active comparator
* pregnant or breast-feeding, or plans to become pregnant at any time during duration of study
* current use of hydroxyurea
* use of noninsulin glucose-lowering medications other than metformin, weight loss medications or dietary supplements for weight loss within 30 days, or anticipated use during the course of the study
* received any investigational drug within prior 30 days
* Clinically significant abnormalities on screening laboratory testing including liver enzymes
* Presence of a medical condition or use of a medication that could compromise the results of the study or the safety of the subject (eg. alcohol or drug abuse, uncontrolled hypertension, history of transient ischemic attack or stroke within the last 12 months)
* employed by or having immediate family members employed by the sponsor or directly involved in conducting the clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
hypoglycemia events | during the first 6 weeks of the maintenance period
  CGM-measured rates of nocturnal level 2 hypoglycemia events
hypoglycemia percentage of time | during the first 6 weeks of maintenance period
  CGM-measured nocturnal percent time

SECONDARY OUTCOMES:
blood chemistry values | baseline through study completion, an average of 7 months
  Triglyceride levels, Liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Weinstock, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (27):
- United States (27):
  - Marvel Clinical Research, Huntington Beach, California
  - Pasadena Clinical Trials, Pasadena, California
  - Diabetes Research Center, Tustin, California
  - University of Colorado, Barbara Davis Center, Denver, Colorado
  - East Coast Institute for Research, Jacksonville, Florida
  - University of Miami Diabetes Research Institute, Miami, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Coast Institute for Research, Canton, Georgia
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - University of Chicago Kovler Diabetes Center, Chicago, Illinois
  - Endeavor Health, Skokie, Illinois
  - Indiana Medical Research Institute, Merrillville, Indiana
  - SUNY Upstate Medical University, Syracuse, New York
  - Asheville Clinical Research, Asheville, North Carolina
  - UNC EnDO Clinical Research Unit, Chapel Hill, North Carolina
  - Physician's East, Greenville, North Carolina
  - University Hospitals Medical Center, Cleveland, Ohio
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Tekton Research, LLC, Irving, Texas
  - Tekton Research, LLC, McKinney, Texas
  - Texas Diabetes % Endocrinology, Round Rock, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Tekton Research, LLC, San Antonio, Texas
  - Wasatch Clinical Research, LLC 310, Salt Lake City, Utah
  - Virginia Endocrinology Research, Chesapeake, Virginia

IPD SHARING:
Plan to Share IPD: No